CLINICAL TRIAL: NCT01707160
Title: A Randomised, Double-blind 2 Way Crossover Trial to Investigate the Pharmacokinetics and Pharmacodynamics of Insulin X14 30/70 PreMix Compared to Human Insulin 30/70 PreMix in Healthy Volunteers
Brief Title: Pharmacokinetics and Pharmacodynamics of Biphasic Insulin Aspart 30 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ANA/DCD/031
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; biphasic human insulin 30

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment period 1 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic human insulin 30
- Treatment period 2 (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic human insulin 30

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — One single dose of each trial drug separated by 4-10 days injected subcutaneously (s.c, under the skin) in random order
Drug: biphasic human insulin 30 — One single dose of each trial drug separated by 4-10 days injected subcutaneously (s.c, under the skin) in random order

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the pharmacokinetics and pharmacodynamics of insulin X14 30/70 PreMix compared to human insulin 30/70 PreMix in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers
* BMI (body mass index) maximum 27 kg/m^2
* HbA1c (glycosylated haemoglobin A1c): 3.4-6.1%
* FBG (fasting blood glucose) maximum 6.0 mmol/L

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 1995-11; Primary Completion 1995-12 (Actual); Study Completion 1995-12 (Actual)

PRIMARY OUTCOMES:
Area under the Curve

SECONDARY OUTCOMES:
Maximum insulin concentration (Cmax)
Time to maximum insulin concentration (tmax)
Minimum glucose concentration (Cmin(glu))
Time to minimum glucose concentration (tmin(glu))
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR,1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Leeds, United Kingdom

REFERENCES:
- [Result] Jacobsen LV, Sogaard B, Riis A. Pharmacokinetics and pharmacodynamics of a premixed formulation of soluble and protamine-retarded insulin aspart. Eur J Clin Pharmacol. 2000 Aug;56(5):399-403. doi: 10.1007/s002280000159. PMID 11009049
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com